CLINICAL TRIAL: NCT00977574
Title: A Three Arm Randomized Phase II Study of Paclitaxel/Carboplatin/Bevacizumab (NSC #704865), Paclitaxel/Carboplatin/Temsirolimus (NSC #683864) and Ixabepilone (NSC #710428)/Carboplatin/Bevacizumab as Initial Therapy for Measurable Stage III or IVA, Stage IVB, or Recurrent Endometrial Cancer
Brief Title: Paclitaxel, Carboplatin, and Bevacizumab or Paclitaxel, Carboplatin, and Temsirolimus or Ixabepilone, Carboplatin, and Bevacizumab in Treating Patients With Stage III, Stage IV, or Recurrent Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01969; NCI-2011-01969 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0086P; CDR0000654472; GOG-0086P (Other: NRG Oncology); GOG-0086P (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-09-12; First posted 2009-09-15 (Estimated); Results first posted 2018-02-27 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Adenosquamous Carcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Recurrent Malignant Uterine Corpus Neoplasm; Stage IIIA Uterine Corpus Carcinoma or Carcinosarcoma by AJCC v7 Stage; Stage IIIB Uterine Corpus Carcinoma or Carcinosarcoma by AJCC v7 Stage; Stage IIIC Uterine Corpus Carcinoma or Carcinosarcoma by AJCC v7 Stage; Stage IVA Uterine Corpus Carcinoma or Carcinosarcoma by AJCC v7 Stage; Stage IVB Uterine Corpus Carcinoma or Carcinosarcoma by AJCC v7 Stage
MeSH Terms: interventions — Bevacizumab; Immunoglobulin G; Disulfides; Carboplatin; ixabepilone; Epothilones; Paclitaxel; Taxes; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (paclitaxel, carboplatin, bevacizumab) (Experimental): Patients receive paclitaxel IV over 3 hours, carboplatin IV over 30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel
- Arm II (paclitaxel, carboplatin, temsirolimus) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and temsirolimus IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Temsirolimus
- Arm III (ixabepilone, carboplatin, bevacizumab) (Experimental): Patients receive ixabepilone IV over 1 hour, carboplatin IV over 30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Drug: Ixabepilone; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm I (paclitaxel, carboplatin, bevacizumab); Arm III (ixabepilone, carboplatin, bevacizumab)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Ixabepilone — Given IV
  Other Names: (1S,3S,7S,10R,11S,12S,16R)-7,11-Dihydroxy-8,8,10,12,16-pentamethyl-3-[(1E)-1-methyl-2-(2-methyl-4-thiazolyl)ethenyl]-17-oxa-4-azabicyclo[14.1.0]heptadecane-5,9-dione; Azaepothilone B; BMS 247550; BMS-247550; BMS247550; Epothilone; Epothilone-B BMS 247550; Ixempra
  Arms: Arm III (ixabepilone, carboplatin, bevacizumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm I (paclitaxel, carboplatin, bevacizumab); Arm II (paclitaxel, carboplatin, temsirolimus)
Drug: Temsirolimus — Given IV
  Other Names: CCI 779; CCI-779; CCI-779 Rapamycin Analog; CCI779; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
  Arms: Arm II (paclitaxel, carboplatin, temsirolimus)

SUMMARY:
This randomized phase II trial studies paclitaxel, carboplatin, and bevacizumab or paclitaxel, carboplatin, and temsirolimus or ixabepilone, carboplatin, and bevacizumab to see how well they work in treating patients with stage III, stage IV, or recurrent endometrial cancer. Drugs used in chemotherapy, such as paclitaxel, carboplatin, and ixabepilone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known which treatment regimen is most effective in treating patients with endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the hazard of progression or death of each of the three arms relative to that of historical controls in patients with advanced or recurrent endometrial cancer.

SECONDARY OBJECTIVES:

I. To determine the nature, frequency, and maximum degree of toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v)3.0 for each of the three arms.

II. To estimate the distribution of the duration of overall survival for each of the three arms.

III. To estimate the proportion of patients with measurable disease who have confirmed objective tumor responses by treatment.

TERTIARY OBJECTIVES:

I. Explore the associations between select biomarkers and progression-free survival as well as secondary measures of clinical outcome (overall survival, tumor response, or disease status if possible) in the context of histologic cell type and treatment.

IA. Somatic mutations in phosphatase and tensin homolog (PTEN)/ phosphoinositide-3-kinase (PI3K) and RAS pathway members by Sequenom mutational profiling and targeted sequencing of candidate genes.

IB. Microsatellite instability by analysis of five National Cancer Institute consensus microsatellite markers (BAT25, BAT26, D2S2123, D5S346, and D17S250) using the Applied Biosystems (ABI) Prism 3100 Genetic Analyzer.

IC. Copy number alterations (gains or losses) by array comparative genomic hybridization (aCGH).

ID. Tumor expression of PTEN and class III beta-tubulin using immunohistochemistry.

IE. Concentration of vascular endothelial growth factor (VEGF) in pre-cycle 1 plasma using an enzyme-linked immunosorbent assay.

II. Explore the relationship among the various biomarkers by histologic subtype and treatment.

III. Explore which combination of biomarkers and clinical covariates optimally predicts responsiveness and resistance to the three treatment arms.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 3 hours, carboplatin IV over 30 minutes, and bevacizumab* IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients undergoing treatment post-surgery (=< 12 weeks) receive bevacizumab beginning on course 2.

ARM II: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and temsirolimus* IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive temsirolimus IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients undergoing treatment post-surgery (=< 12 weeks) receive temsirolimus beginning on course 2.

ARM III: Patients receive ixabepilone IV over 1 hour, carboplatin IV over 30 minutes, and bevacizumab* IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients undergoing treatment post-surgery (=< 12 weeks) receive bevacizumab beginning on course 2.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable stage III, measurable stage IVA, stage IVB (with or without measurable disease) or recurrent (with or without measurable disease) endometrial carcinoma

  * Histologic confirmation of the original primary tumor is required; patients with the following histologic epithelial cell types are eligible: endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell carcinoma, and transitional cell carcinoma
* Measurable disease is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1); measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have Gynecologic Oncology Group (GOG) performance status of 0, 1, or 2
* Patients must not be eligible for a higher priority GOG protocol, if one exists; in general, this would refer to any active GOG Phase III protocol or Rare Tumor protocol for the same patient population
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl equivalent to Common Terminology Criteria (CTCAE v3.0) grade 1
* Platelets greater than or equal to 100,000/mcl
* Creatinine less than or equal to 1.5 times institutional upper limit normal (ULN), CTCAE v3.0 grade 1
* Bilirubin less than or equal to 1.5 x ULN (CTCAE v3.0 grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) less than or equal to 2.5 x ULN (CTCAE v3.0 grade 1)
* Alkaline phosphatase less than or equal to 2.5 x ULN (CTCAE v3.0 grade 1)
* Urine protein creatinine (UPC) ratio must be < 1.0 gram (gm); if UPC ratio >= 1, collection of 24-hour urine measurement of urine protein is recommended (24-hour urine protein level must be < 1000 mg for patient enrollment)

  * UPC ratio of spot urine is an estimation of the 24 urine protein excretion

    * A UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) =< 1.5 x ULN
* Fasting cholesterol less than 300 mg/dL (CTCAE v3.0 grade 1)
* Fasting triglycerides =< 2.5 x ULN (CTCAE v3.0 grade 1)
* Patients must NOT have received prior chemotherapy or targeted therapy, including chemotherapy used for radiation sensitization for treatment of endometrial carcinoma
* Patients must NOT have received prior therapy with bevacizumab or other VEGF pathway targeted therapy; patients must NOT have received prior therapy with temsirolimus, everolimus, ridaforolimus, sirolimus, or any other PI3K/ v-akt murine thymoma viral oncogene homolog 1 (AKT)/mammalian target of rapamycins (mTor) pathway targeted therapy
* Patients may have receive prior radiation therapy for treatment of endometrial carcinoma; prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para-aortic radiation therapy, and/or intravaginal brachytherapy; all radiation therapy must be completed at least 4 weeks prior to the first date of study therapy; the prior radiation field, radiation dose, number of fractions and prior radiation start and stop dates must be provided on the Fast Fact Sheet (FFS) at registration
* Patients may have received prior hormonal therapy for treatment of endometrial carcinoma; all hormonal therapy must be discontinued at least one week prior to the first date of study therapy
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, and other specific malignancies as noted below, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of endometrial cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with serious, non-healing wound, ulcer, or bone fracture; this includes history of abdominal/pelvic fistula, gastrointestinal perforation or intra-abdominal abscess within 3 months prior to the first date of study therapy; patients with underlying lesions that caused the fistula or perforation in the past that have not been corrected
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy or any brain metastases
* Patients with clinically significant cardiovascular disease; this includes:

  * Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg
  * Myocardial infarction or unstable angina within 6 months of the first date of study therapy
  * New York Heart Association (NYHA) class II or greater congestive heart failure
  * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication)
  * CTCAE grade 2 or greater peripheral vascular disease.
  * History of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of study therapy.
  * Aortic aneurysm and/or history of aortic dissection
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Patients undergoing invasive procedures as defined below:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of bevacizumab or temsirolimus therapy
  * Major surgical procedure anticipated during the course of the study.
  * Minor surgical procedures, fine needle aspirates, or core biopsies within 7 days prior to the first date of study therapy
* Patients with known prior history of interstitial pneumonitis
* Patients with CTCAE v. 3, grade 2 or greater hypoxemia
* Patients with CTCAE v. 3, grade 2 or greater dyspnea
* Patients must not have uncontrolled diabetes, and must not have baseline hemoglobin A1C (HgbA1C) > 8
* Patients with peripheral neuropathy > CTCAE v.3, grade 1
* Patients who are pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2009-09-14 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2026-03-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Aghajanian, Principal Investigator — NRG Oncology
Locations (230):
- United States (230):
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - John Muir Medical Center-Concord, Concord, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - San Diego VA Medical Center, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Gynecologic Oncology PC, Englewood, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Saint Luke's Hospital-Warren Campus, Phillipsburg, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Hospital Medical Center of Queens, Fresh Meadows, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Oncology Associates PA, Columbia, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

REFERENCES:
- [Derived] Thiel KW, Devor EJ, Filiaci VL, Mutch D, Moxley K, Alvarez Secord A, Tewari KS, McDonald ME, Mathews C, Cosgrove C, Dewdney S, Aghajanian C, Samuelson MI, Lankes HA, Soslow RA, Leslie KK. TP53 Sequencing and p53 Immunohistochemistry Predict Outcomes When Bevacizumab Is Added to Frontline Chemotherapy in Endometrial Cancer: An NRG Oncology/Gynecologic Oncology Group Study. J Clin Oncol. 2022 Oct 1;40(28):3289-3300. doi: 10.1200/JCO.21.02506. Epub 2022 Jun 3. PMID 35658479
- [Derived] Leslie KK, Filiaci VL, Mallen AR, Thiel KW, Devor EJ, Moxley K, Richardson D, Mutch D, Secord AA, Tewari KS, McDonald ME, Mathews C, Cosgrove C, Dewdney S, Casablanca Y, Jackson A, Rose PG, Zhou X, McHale M, Lankes H, Levine DA, Aghajanian C. Mutated p53 portends improvement in outcomes when bevacizumab is combined with chemotherapy in advanced/recurrent endometrial cancer: An NRG Oncology study. Gynecol Oncol. 2021 Apr;161(1):113-121. doi: 10.1016/j.ygyno.2021.01.025. Epub 2021 Feb 2. PMID 33541735

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual of 349 patients from 48 main members and CCOP sites began on 9/14/2009 and completed on 01/09/2012 in 28 months; 5 months longer than expected. There were 11 patients deemed ineligible by central review most for reasons related to pathologic diagnosis. Ten patients refused all protocol treatment.
Groups:
- Arm I (Paclitaxel, Carboplatin, Bevacizumab): Paclitaxel 175 mg/m2 IV over 3 hours day 1 Carboplatin AUC = 6 IV day 1 Bevacizumab 15mg/kg IV day 1 (starting with cycle 2 for those patients who are entering post surgery) Maintenance regimen - Bevacizumab 15mg/kg IV every 21 days
- Arm II (Paclitaxel, Carboplatin, Temsirolimus): Paclitaxel 175 mg/m2 IV over 3 hours day 1 Carboplatin AUC = 5 IV day 1 Temsirolimus 25 mg IV days 1 and 8 (starting with cycle 2 for those patients who are entering post surgery) Maintenance regimen - Temsirolimus 25 mg IV weekly days 1, 8 and 15 (one cycle = 21 days)
- Arm III (Ixabepilone, Carboplatin, Bevacizumab): Ixabepilone 30 mg/m2 IV over 1 hour day 1 Carboplatin AUC = 6 IV day 1 Bevacizumab 15mg/kg IV day 1 (starting with cycle 2 for those patients who are entering post surgery) Maintenance regimen - Bevacizumab 15mg/kg IV every 21 days
Period: Overall Study
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevacizumab) | Arm II (Paclitaxel, Carboplatin, Temsirolimus) | Arm III (Ixabepilone, Carboplatin, Bevacizumab)
Started | 116 | 115 | 118
Completed | 112 | 113 | 114
Not Completed | 4 | 2 | 4
Not completed — Never Treated | 4 | 2 | 4

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevacizumab) | Arm II (Paclitaxel, Carboplatin, Temsirolimus) | Arm III (Ixabepilone, Carboplatin, Bevacizumab) | Total
Number analyzed (Participants) | 116 | 115 | 118 | 349
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 2 | 2 | 3 | 7
  40-49 years | 6 | 5 | 8 | 19
  50-59 years | 36 | 35 | 19 | 90
  60-69 years | 48 | 50 | 57 | 155
  70-79 years | 22 | 22 | 28 | 72
  >=80 years | 2 | 1 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 115 | 118 | 349
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Progressed or Died by 25 Months From Enrollment
Description: PFS (Progression free survival) is defined as the duration of time from date of study entry to time of progression or death, whichever occurs first. Patients with a status of alive, progression-free are censored at their date of last follow-up. To lessen the potential for bias in the progression evaluation times between treatment arms and historical controls, progression/death times will be grouped over 6 18-week time intervals. Progressions are carried forward to the end of the interval. All progressions or deaths occurring after the 6th 18-week interval are censored at 25 months for this analysis. Study NCT00977574
Time Frame: at 25 months
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevacizumab) | Arm II (Paclitaxel, Carboplatin, Temsirolimus) | Arm III (Ixabepilone, Carboplatin, Bevacizumab)
Number analyzed (Participants) | 116 | 115 | 118
Participants | 86 | 96 | 88

2. Secondary Outcome: Frequency and Severity of Toxicity as Assessed by CTCAE v3.0 for Each of the Three Arms.
Time Frame: Median of 10 cycles of treatment plus 30 days
Population: Treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevacizumab) | Arm II (Paclitaxel, Carboplatin, Temsirolimus) | Arm III (Ixabepilone, Carboplatin, Bevacizumab)
Number analyzed (Participants) | 112 | 113 | 114
Participants
  Any Adverse Event, Any Grade | 112 | 113 | 114
  Any Adverse Event, Grades >= 3 | 105 | 111 | 109
  Any Adverse Event, Grade 5 | 4 | 6 | 6

3. Secondary Outcome: The Median Duration of Overall Survival for Each of the Three Arms.
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Time from date of study entry to time of death or the date of last contact, assessed up to 5 years
Population: All enrolled patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevacizumab) | Arm II (Paclitaxel, Carboplatin, Temsirolimus) | Arm III (Ixabepilone, Carboplatin, Bevacizumab)
Number analyzed (Participants) | 116 | 115 | 118
months | 34 [26.0 to 51.4] | 25 [18.5 to 29.6] | 25.2 [18.8 to 32.1]

4. Secondary Outcome: The Proportion of Patients With Measurable Disease Who Have Confirmed Objective Tumor Responses by Treatment.
Description: RECIST 1.1 was used to define objective tumor response. A complete response is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. A partial response is defined as At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. There can be no unequivocal progression of non-target lesions and no new lesions. Complete and partial responses are included in the objective tumor response rate. Confirmation of response was not required.
Time Frame: Imaging was done every 3 cycles and at any other time clinically indicated. Imaging was required every 9 weeks until progression or initiation on non protocol therapy. After 2 years of protocol therapy or follow up, CT scan or MRI was every 3 months
Population: Enrolled patients with measurable disease
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevacizumab) | Arm II (Paclitaxel, Carboplatin, Temsirolimus) | Arm III (Ixabepilone, Carboplatin, Bevacizumab)
Number analyzed (Participants) | 89 | 85 | 85
Participants | 53 | 47 | 45

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Arm/Group | Arm I (Paclitaxel, Carboplatin, Bevacizumab) | Arm II (Paclitaxel, Carboplatin, Temsirolimus) | Arm III (Ixabepilone, Carboplatin, Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 48/112 | 57/113 | 53/114
Other Adverse Events (participants affected / at risk) | 112/112 | 113/113 | 113/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel, Carboplatin, Bevacizumab) (N=112) | Arm II (Paclitaxel, Carboplatin, Temsirolimus) (N=113) | Arm III (Ixabepilone, Carboplatin, Bevacizumab) (N=114)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Neutrophils (Blood and lymphatic system disorders) | 2 | 4 | 1
Platelets (Blood and lymphatic system disorders) | 3 | 1 | 4
Leukocytes (Blood and lymphatic system disorders) | 0 | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 4 | 1 | 1
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 1
Vasovagal Episode (Cardiac disorders) | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac Ischemia/Infarction (Cardiac disorders) | 1 | 0 | 1
Hypertension (Cardiac disorders) | 0 | 0 | 1
Left Venticular Diastolic Dysfunction (Cardiac disorders) | 0 | 0 | 1
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 1 | 0
Inr (Vascular disorders) | 0 | 1 | 0
Fever (General disorders) | 0 | 1 | 1
Weight Loss (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2
Death No Ctcae Term - Disease Progression Nos (General disorders) | 0 | 1 | 0
Death No Ctcae Term - Death Nos (General disorders) | 2 | 1 | 4
Death No Ctcae Term - Multi-Organ Failure (General disorders) | 0 | 0 | 1
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Fistula, Gi - Colon/Cecum/Appendix (Gastrointestinal disorders) | 0 | 0 | 1
Perforation, Gi - Colon (Gastrointestinal disorders) | 1 | 1 | 0
Fistula, Gi - Rectum (Gastrointestinal disorders) | 1 | 0 | 1
Obstruction, Gi - Colon (Gastrointestinal disorders) | 2 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Leak, Gi - Small Bowel (Gastrointestinal disorders) | 0 | 0 | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Perforation, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3
Dehydration (Gastrointestinal disorders) | 2 | 1 | 5
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 0 | 0 | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 0 | 0 | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 1 | 0 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0
Hemorrhage/Pulmonary - Bronchus (Vascular disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 2 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Soft Tissue Nos (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bone (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 0 | 2 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 1 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 1 | 2 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 2 | 2 | 0
Febrile Neutropenia (Infections and infestations) | 2 | 2 | 2
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 0 | 2 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 0 | 0 | 2
Inf Unknown Anc: Blood (Infections and infestations) | 2 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Bladder (Urinary) (Infections and infestations) | 0 | 0 | 1
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Nerve-Peripheral (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Pharynx (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 1 | 0 | 1
Inf Unknown Anc: Wound (Infections and infestations) | 0 | 2 | 0
Inf Unknown Anc: Foreign Body (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Foreign Body (Infections and infestations) | 0 | 2 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Catheter-Related (Infections and infestations) | 1 | 1 | 0
Edema: Limb (Blood and lymphatic system disorders) | 0 | 1 | 0
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1 | 0 | 0
Proteinuria (Metabolism and nutrition disorders) | 2 | 0 | 2
Creatinine (Metabolism and nutrition disorders) | 1 | 0 | 0
Alkaline Phosphatase (Metabolism and nutrition disorders) | 0 | 0 | 1
Bilirubin (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Soft Tissue Necrosis - Abdomen (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 3 | 0 | 0
Neurology - Other (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1
Cns Ischemia (Nervous system disorders) | 1 | 0 | 0
Confusion (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Neuropathy-Motor (Nervous system disorders) | 1 | 0 | 0
Pain: Chest /Thorax Nos (General disorders) | 0 | 2 | 0
Pain: Head/Headache (General disorders) | 1 | 0 | 2
Pain: Back (General disorders) | 0 | 2 | 0
Pain: Joint (General disorders) | 0 | 0 | 1
Pain: Gallbladder (General disorders) | 0 | 0 | 1
Pain: Abdominal Pain Nos (General disorders) | 2 | 1 | 3
Pain: Muscle (General disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0
Obstruction, Gu - Ureter (Renal and urinary disorders) | 0 | 0 | 1
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 1 | 1 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 4 | 4 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Paclitaxel, Carboplatin, Bevacizumab) (N=112) | Arm II (Paclitaxel, Carboplatin, Temsirolimus) (N=113) | Arm III (Ixabepilone, Carboplatin, Bevacizumab) (N=114)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 6 | 5 | 13
Rhinitis (Immune system disorders) | 24 | 15 | 20
Otitis Middle Ear (Ear and labyrinth disorders) | 2 | 0 | 0
Auditory/Ear - Other (Ear and labyrinth disorders) | 3 | 3 | 3
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 6 | 3 | 6
Tinnitus (Ear and labyrinth disorders) | 13 | 6 | 12
Hearing (Monitoring Program) (Ear and labyrinth disorders) | 0 | 0 | 3
Neutrophils (Blood and lymphatic system disorders) | 106 | 106 | 102
Platelets (Blood and lymphatic system disorders) | 87 | 96 | 101
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 | 0 | 2
Leukocytes (Blood and lymphatic system disorders) | 110 | 110 | 105
Lymphopenia (Blood and lymphatic system disorders) | 9 | 8 | 6
Hemoglobin (Blood and lymphatic system disorders) | 105 | 111 | 110
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1 | 4 | 0
Palpitations (Cardiac disorders) | 5 | 5 | 4
Cardiac Arrhythmia - Other (Cardiac disorders) | 0 | 0 | 1
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 5 | 1 | 3
Vasovagal Episode (Cardiac disorders) | 1 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 1
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 2 | 0 | 2
Ventricular Arrhythmia - Arrhythmia Nos (Cardiac disorders) | 1 | 0 | 0
Ventricular Arrhythmia - Pvcs (Cardiac disorders) | 1 | 0 | 0
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 | 1 | 0
Hypertension (Cardiac disorders) | 51 | 18 | 50
Valvular Heart Disease (Cardiac disorders) | 1 | 0 | 0
Left Venticular Diastolic Dysfunction (Cardiac disorders) | 0 | 0 | 1
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 0 | 1
Hypotension (Cardiac disorders) | 6 | 3 | 5
Cardipulmonary Arrest (Cardiac disorders) | 0 | 0 | 1
Inr (Vascular disorders) | 4 | 9 | 8
Coagulopathy - Other (Vascular disorders) | 1 | 1 | 1
Ptt (Vascular disorders) | 4 | 4 | 5
Constitutional Symptoms - Other (General disorders) | 5 | 0 | 4
Sweating (General disorders) | 4 | 0 | 3
Weight Gain (General disorders) | 16 | 7 | 8
Patient Odor (General disorders) | 0 | 1 | 0
Fever (General disorders) | 17 | 14 | 14
Weight Loss (General disorders) | 24 | 29 | 31
Hypothermia (General disorders) | 1 | 0 | 1
Rigors/Chills (General disorders) | 6 | 4 | 7
Fatigue (General disorders) | 100 | 90 | 98
Insomnia (General disorders) | 24 | 31 | 22
Death No Ctcae Term - Disease Progression Nos (General disorders) | 0 | 0 | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 10 | 17 | 8
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 88 | 81 | 83
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cheilitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Bruising (Skin and subcutaneous tissue disorders) | 10 | 9 | 9
Acne (Skin and subcutaneous tissue disorders) | 2 | 10 | 1
Rash (Skin and subcutaneous tissue disorders) | 18 | 52 | 19
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 10 | 3
Decubitus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Atrophy, Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 18 | 12
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Flushing (Skin and subcutaneous tissue disorders) | 5 | 11 | 6
Hand-Foot (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 5 | 8 | 3
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Ulceration (Skin and subcutaneous tissue disorders) | 2 | 4 | 3
Hot Flashes (Endocrine disorders) | 12 | 9 | 5
Endocrine - Other (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0
Salivary Gland Changes (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 4 | 2 | 4
Fistula, Gi - Rectum (Gastrointestinal disorders) | 0 | 0 | 1
Obstruction, Gi - Colon (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 2 | 0 | 2
Hemorrhoids (Gastrointestinal disorders) | 5 | 2 | 3
Heartburn (Gastrointestinal disorders) | 12 | 7 | 8
Mucositis (Functional/Sympt) - Esophagus (Gastrointestinal disorders) | 0 | 1 | 0
Dental: Teeth (Gastrointestinal disorders) | 2 | 0 | 0
Leak, Gi - Leak Nos (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 4 | 2
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 7 | 6 | 9
Distention (Gastrointestinal disorders) | 5 | 6 | 8
Taste Alteration (Gastrointestinal disorders) | 13 | 25 | 17
Incontinence, Anal (Gastrointestinal disorders) | 0 | 1 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 5 | 3
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 14 | 26 | 14
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 3 | 1
Fistula, Gi - Oral Cavity (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0
Mucositis (Clinical Exam) - Stomach (Gastrointestinal disorders) | 1 | 1 | 0
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 15 | 27 | 7
Vomiting (Gastrointestinal disorders) | 46 | 36 | 51
Anorexia (Gastrointestinal disorders) | 53 | 46 | 50
Dehydration (Gastrointestinal disorders) | 13 | 10 | 17
Constipation (Gastrointestinal disorders) | 66 | 58 | 66
Nausea (Gastrointestinal disorders) | 78 | 73 | 81
Gastrointestinal - Other (Gastrointestinal disorders) | 4 | 2 | 3
Diarrhea (Gastrointestinal disorders) | 55 | 47 | 55
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 3 | 1 | 3
Hemorrhage, Gu - Vagina (Vascular disorders) | 11 | 8 | 14
Hemorrhage/Pulmonary - Bronchopulmonary Nos (Vascular disorders) | 0 | 0 | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 5 | 1 | 8
Hemorrhage/Pulmonary - Respiratory Tract Nos (Vascular disorders) | 1 | 0 | 1
Hemorrhage, Gi - Varices (Rectal) (Vascular disorders) | 2 | 0 | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 34 | 24 | 32
Hematoma (Vascular disorders) | 4 | 0 | 2
Hemorrhage, Gi - Anus (Vascular disorders) | 0 | 1 | 1
Hemorrhage, Gu - Uterus (Vascular disorders) | 0 | 0 | 1
Hemorrhage, Gu - Ureter (Vascular disorders) | 0 | 0 | 1
Hemorrhage, Gi - Lower Gi Nos (Vascular disorders) | 1 | 1 | 0
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 3 | 0 | 3
Hemorrhage, Gu - Bladder (Vascular disorders) | 1 | 0 | 1
Petechiae (Vascular disorders) | 1 | 0 | 1
Hemorrhage/Bleeding - Other (Vascular disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Liver Dysfunction (Hepatobiliary disorders) | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Wound (Infections and infestations) | 0 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Dental-Tooth (Infections and infestations) | 2 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Skin (Cellulitis) (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Vulva (Infections and infestations) | 0 | 0 | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 5 | 3 | 9
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 2 | 2 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Eye Nos (Infections and infestations) | 0 | 1 | 0
Inf W/Gr 3 Or 4 Anc: Peritoneal Cavity (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 1 | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 2 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Otitis Media Nos (Infections and infestations) | 2 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 4 | 5 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Heart (Infections and infestations) | 0 | 1 | 0
Febrile Neutropenia (Infections and infestations) | 2 | 2 | 5
Inf W/Nml Or Gr 1 Or 2 Anc: Lip/Perioral (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 1 | 1 | 0
Inf Unknown Anc: Sinus (Infections and infestations) | 0 | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Dental-Tooth (Infections and infestations) | 3 | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 20 | 11 | 17
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 0 | 1 | 1
Inf Unknown Anc: Blood (Infections and infestations) | 0 | 1 | 1
Infection - Other (Infections and infestations) | 8 | 3 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Muscle (Infections and infestations) | 0 | 0 | 1
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 0 | 1 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Conjunctiva (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Vulva (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 0 | 2 | 2
Inf W/Gr 3 Or 4 Anc: Abdomen Nos (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 1 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Pharynx (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 2 | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 3 | 2 | 4
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 0 | 0 | 1
Inf Unknown Anc: Eye Nos (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Lymphatic (Infections and infestations) | 0 | 1 | 0
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 5 | 2 | 2
Inf Unknown Anc: Catheter-Related (Infections and infestations) | 0 | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Foreign Body (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Vagina (Infections and infestations) | 1 | 0 | 0
Inf W/Gr 3 Or 4 Anc: Upper Airway Nos (Infections and infestations) | 0 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Sinus (Infections and infestations) | 2 | 0 | 1
Inf W/Gr 3 Or 4 Anc: Nerve-Peripheral (Infections and infestations) | 1 | 0 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 1 | 0 | 0
Inf Unknown Anc: Ungual (Nails) (Infections and infestations) | 0 | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 2 | 1 | 3
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 4 | 2 | 6
Inf W/Gr 3 Or 4 Anc: Catheter-Related (Infections and infestations) | 1 | 1 | 0
Lymphatics - Other (Blood and lymphatic system disorders) | 0 | 1 | 0
Edema: Viscera (Blood and lymphatic system disorders) | 0 | 0 | 1
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 0 | 3 | 0
Edema: Limb (Blood and lymphatic system disorders) | 25 | 46 | 28
Edema: Head And Neck (Blood and lymphatic system disorders) | 1 | 6 | 3
Ast (Metabolism and nutrition disorders) | 20 | 26 | 20
Gfr (Metabolism and nutrition disorders) | 1 | 2 | 3
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 5 | 7 | 8
Alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Cholesterol,serum High (Metabolism and nutrition disorders) | 7 | 35 | 2
Proteinuria (Metabolism and nutrition disorders) | 16 | 1 | 15
Creatinine (Metabolism and nutrition disorders) | 21 | 21 | 21
Hypoalbuminemia (Metabolism and nutrition disorders) | 23 | 31 | 28
Alt (Metabolism and nutrition disorders) | 21 | 21 | 16
Alkaline Phosphatase (Metabolism and nutrition disorders) | 19 | 25 | 20
Bilirubin (Metabolism and nutrition disorders) | 7 | 7 | 9
Hypermagnesemia (Metabolism and nutrition disorders) | 7 | 3 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 13 | 20 | 9
Hyponatremia (Metabolism and nutrition disorders) | 27 | 24 | 34
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 | 31 | 5
Cpk (Metabolism and nutrition disorders) | 0 | 1 | 0
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 4 | 4 | 3
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 5 | 4 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 21 | 28 | 30
Hyperkalemia (Metabolism and nutrition disorders) | 12 | 8 | 10
Hyperglycemia (Metabolism and nutrition disorders) | 44 | 48 | 38
Hypokalemia (Metabolism and nutrition disorders) | 27 | 43 | 30
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 4 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 7 | 4 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 45 | 36 | 33
Seroma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 7 | 0 | 4
Joint-Function (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3
Fracture (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2
Extremity-Upper (Function) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gait/Walking (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 9 | 3 | 8
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 13 | 11 | 12
Muscle Weakness - Trunk (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4
Syncope (Nervous system disorders) | 5 | 3 | 4
Involuntary Movement (Nervous system disorders) | 1 | 1 | 2
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Neurology - Other (Nervous system disorders) | 3 | 2 | 1
Mental Status (Nervous system disorders) | 0 | 0 | 1
Mood Alteration - Depression (Nervous system disorders) | 19 | 17 | 19
Mood Alteration - Anxiety (Nervous system disorders) | 16 | 17 | 19
Mood Alteration - Agitation (Nervous system disorders) | 1 | 1 | 1
Tremor (Nervous system disorders) | 2 | 1 | 3
Speech Impairment (Nervous system disorders) | 2 | 1 | 2
Seizure (Nervous system disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Cognitive Disturbance (Nervous system disorders) | 5 | 0 | 0
Confusion (Nervous system disorders) | 4 | 1 | 4
Memory Impairment (Nervous system disorders) | 6 | 5 | 4
Dizziness (Nervous system disorders) | 31 | 12 | 27
Neuropathy,cranial - Cn Viii Hearing/Balance (Nervous system disorders) | 0 | 0 | 1
Neuropathy,cranial - Cn I Smell (Nervous system disorders) | 0 | 1 | 0
Neuropathy-Sensory (Nervous system disorders) | 79 | 77 | 69
Neuropathy-Motor (Nervous system disorders) | 11 | 4 | 6
Ocular/Visual - Other (Eye disorders) | 7 | 1 | 1
Uveitis (Eye disorders) | 0 | 0 | 1
Proptosis/Enophthalmos (Eye disorders) | 1 | 0 | 0
Watery Eye (Eye disorders) | 0 | 4 | 2
Glaucoma (Eye disorders) | 0 | 0 | 1
Dry Eye (Eye disorders) | 1 | 3 | 3
Ocular Surface Disease (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 2 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 1
Flashing Lights/Floaters (Eye disorders) | 4 | 2 | 6
Diplopia (Eye disorders) | 0 | 0 | 2
Blurred Vision (Eye disorders) | 19 | 10 | 20
Eyelid Dysfunction (Eye disorders) | 1 | 0 | 0
Pain - Other (General disorders) | 9 | 6 | 12
Pain: Urethra (General disorders) | 4 | 3 | 1
Pain: Pelvis (General disorders) | 6 | 4 | 2
Pain: Breast (General disorders) | 0 | 1 | 1
Pain: Vagina (General disorders) | 3 | 2 | 1
Pain: Chest /Thorax Nos (General disorders) | 9 | 5 | 14
Pain: Chest Wall (General disorders) | 7 | 1 | 3
Pain: Throat/Pharynx/Larynx (General disorders) | 8 | 7 | 4
Pain: Pleura (General disorders) | 0 | 1 | 0
Pain: Eye (General disorders) | 0 | 1 | 0
Pain: Head/Headache (General disorders) | 51 | 21 | 39
Pain: Neck (General disorders) | 6 | 3 | 4
Pain: Extremity-Limb (General disorders) | 39 | 23 | 29
Pain: Buttock (General disorders) | 0 | 3 | 0
Pain: Back (General disorders) | 27 | 19 | 20
Pain: Joint (General disorders) | 52 | 30 | 42
Pain: Bone (General disorders) | 8 | 5 | 12
Pain: Kidney (General disorders) | 0 | 0 | 1
Pain: Bladder (General disorders) | 3 | 0 | 4
Pain: Pain Nos (General disorders) | 7 | 4 | 6
Pain: Stomach (General disorders) | 3 | 0 | 0
Pain: Rectum (General disorders) | 3 | 3 | 2
Pain: Oral Cavity (General disorders) | 5 | 8 | 2
Pain: Esophagus (General disorders) | 1 | 0 | 0
Pain: Dental/Teeth/Peridontal (General disorders) | 3 | 1 | 2
Pain: Abdominal Pain Nos (General disorders) | 37 | 40 | 40
Pain: Scalp (General disorders) | 0 | 1 | 3
Pain: Oral - Gums (General disorders) | 3 | 1 | 2
Pain: Skin (General disorders) | 1 | 1 | 1
Pain: Lip (General disorders) | 0 | 1 | 0
Pain: Middle Ear (General disorders) | 2 | 1 | 1
Pain: External Ear (General disorders) | 2 | 1 | 1
Pain: Cardiac/ Heart (General disorders) | 3 | 0 | 1
Pain: Tumor (General disorders) | 0 | 0 | 1
Pain: Muscle (General disorders) | 30 | 37 | 25
Pain: Anus (General disorders) | 1 | 0 | 1
Pain: Neuralgia (General disorders) | 1 | 2 | 2
Pain: Sinus (General disorders) | 3 | 0 | 3
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 7
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 14 | 5 | 12
Edema, Larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 9 | 1 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 48 | 37 | 29
Dlco (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 49 | 39 | 56
Renal/Genitourinary - Other (Renal and urinary disorders) | 5 | 2 | 4
Leak, Gu - Urethra (Renal and urinary disorders) | 0 | 0 | 1
Cystitis (Renal and urinary disorders) | 2 | 1 | 2
Urinary Retention (Renal and urinary disorders) | 3 | 5 | 1
Obstruction, Gu - Urethra (Renal and urinary disorders) | 1 | 0 | 0
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1 | 0 | 1
Incontinence, Urinary (Renal and urinary disorders) | 8 | 8 | 7
Fistula, Gu - Vagina (Renal and urinary disorders) | 2 | 0 | 2
Renal Failure (Renal and urinary disorders) | 1 | 1 | 0
Urinary Frequency (Renal and urinary disorders) | 21 | 16 | 14
Libido (Reproductive system and breast disorders) | 1 | 0 | 0
Irregular Menses (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal Dryness (Reproductive system and breast disorders) | 0 | 2 | 0
Sexual/Reproductive Function: Other (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginitis (Reproductive system and breast disorders) | 0 | 3 | 2
Vaginal Stenosis (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal Mucositis (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 6 | 5 | 4
Syndromes - Other (General disorders) | 1 | 0 | 1
Cytokine Release Syndrome (General disorders) | 1 | 0 | 0
Flu-Like Syndrome (General disorders) | 0 | 1 | 0
Vascular - Other (Vascular disorders) | 0 | 0 | 1
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 1 | 0 | 0
Thrombosis/Thrombus/Embolism (Vascular disorders) | 5 | 10 | 10
Phlebitis (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less